CLINICAL TRIAL: NCT00844259
Title: Functional Communicative Profile of Children With Down Syndrome
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Suelly Cecilia Olivan Limongi, University of Sao Paulo
Other Study IDs: 180875
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Down Syndrome
Keywords: Down syndrome; Pragmatics; Language Development
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Research Group: 15 children with Down syndrome, observed in two interaction conditions: playing with their therapist (A) and playing with their caregiver (B).

SUMMARY:
The aim of this study was to verify the use of communicative functions by children with DS in two interaction conditions: interaction with therapist and interaction with parent.

DETAILED DESCRIPTION:
Parents and caregivers' engagement on therapeutic process of children with Down syndrome (DS) is important for language and communication development. The identification of the communicative skills presented by these children as well as the context influence in their performance as interlocutors, will contribute to the design of therapeutic interventions.

Pragmatics theories are helpful to language use studies, since it takes into account social and environmental aspects and considers adult-child interaction as a determinant factor for its occurrence.

ELIGIBILITY:
Inclusion Criteria:

* genetic diagnosis of Down syndrome
* good health conditions
* normal results on audiologic evaluation
* pediatric and ear, nose and throat periodic check ups.
* attend speech-language therapy at the Speech Language Pathology Laboratory in Syndromes and Sensorimotor Deficits (SLPL-SSD) of the School of Medicine of the University of São Paulo.

Exclusion Criteria:

* submission to long term hospitalizations due to heart diseases and major respiratory airway infections, that may interfere in the child's global development
* presence of visual or auditory important deficits

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 15 children with Down syndrome aged from 5 to 8 years.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2006-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suelly CO Limongi, PhD, Study Chair — University of Sao Paulo; Eliza P Cunha, Ms student, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo - School of Medicine - Department of Physiotherapy, Communication Sciences and Disorders, Occupational Therapy, São Paulo, São Paulo, Brazil